CLINICAL TRIAL: NCT01509443
Title: Application of Breathing Exercise Program to Improve Asthma in Obese Patients: Effects on Clinico-immunological Parameters
Brief Title: Breathing & Mild Physical Exercise Therapy for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Rasheed Ahmad, PhD, Principal Investigator, Dasman Diabetes Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RA-2011-015
Record Dates: First submitted 2012-01-02; First posted 2012-01-13 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: Asthma; Obesity; Breathing exercise
MeSH Terms: conditions — Asthma; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Experimental): Participants will receive standard asthmatic treatment and breathing/mild physical exercise
  Interventions: Other: Exercise
- Control Arm (No Intervention): The control arm will receive standard medical care for asthma

INTERVENTIONS:
Other: Exercise — Participants will perform 2-4 sessions of the prescribed exercise every day (One session: deep breathing 5-10 times; upper body stretching 5-10 times).
  Other Names: Deep breathing and mild physical exercise
  Arms: Interventional

SUMMARY:
Overall goal: To apply the investigators' well defined simple, few-minute breathing/ mild physical exercise program and evaluate its efficacy/benefits for the improvement of clinico-immunological outcome in obese patients with asthma.

Rationale & Hypothesis: Different breathing exercise regimens currently recommended are not well defined and in certain cases may worsen dyspnea or even trigger an asthma attack. Therefore, it is important to evaluate the overall usefulness of a breathing exercise as a therapeutic intervention of asthma. In this regard, the investigators have designed an easy, few-minute breathing exercise program as a treatment modality for asthma and to evaluate its efficacy in improving associated clinico-immunological symptoms. The investigators hypothesize that the investigators' well-designed breathing/mild physical exercise intervention for obese patients will help alleviate the stress and symptoms of asthma by reducing the chronic low-grade systemic inflammation and thus potentiate the beneficial outcome of medication to render a better control over the disease and to improve the quality of life in obese patients.

Clinical relevance/Significance:

The investigators expect that their exercise module will help reduce inflammation caused by asthma, and thereby relieving symptoms of asthma. If successful, this would allow regular individualized exercise module to be recommended as a part of therapy for people with asthma, which could possibly reduce the dosage as well as frequency of taking medicine that they need.

DETAILED DESCRIPTION:
Asthmatics particularly obese have major constraints impeding regular physical activity and exercise. Indeed, the few studies that have resorted to the option of exercise in asthmatic patients also recognized the exacerbation of associated symptoms as a major limitation of this approach. Considering the other obstacles that are often involved, such as lack of time and motivation, inadequate social support and lack of access to facilities etc, it is therefore all the more necessary to design a simple, feasible and carefully tailored breathing exercise modality in obese patients with asthma, and to study its impact on the improvement of clinico-immunological parameters, lung function and overall quality of life. To this end, investigators have developed a safe and feasible light breathing exercise program for individuals with asthma based on our previous observations.

Study Aims & Objectives:

The investigators' main goal is to apply a well defined simple exercise program that includes physical and breathing exercise lessons and evaluate its effects on the improvement of clinico-immunological outcome in obese patients with asthma. There are three main objectives based on clinic-immunological outcome.

1. To assess the improvement of asthma control, lung function and airways hyper-reactivity after the intervention.
2. To test if the proposed intervention will result in the improvement of pro-inflammatory profiles.
3. To determine if physical and psychological performances as well as health related quality of life are positively impacted by the proposed exercise modality.

About 200 individuals with asthma will be enrolled in this study and divided into two groups: The intervention group and controls. The intervention group will receive standard asthma care along with breathing/mild physical exercise. The control group will be the asthmatic patients who are not willing to receive the exercise intervention. At study entry, participants will undergo a clinical assessment which includes physical exam, asthma control/ quality of life questionnaires, pulmonary function tests, and lung inflammation test (Exhaled Nitric Oxide). To monitor participants throughout the study, follow up visits will be done at 6, 12, 18 and 24 weeks after starting the exercise. About 40 ml blood will be collected at baseline (pre-exercise) and two different time points (3 and 6 months of post-exercise). The blood samples will be used for pro-inflammatory profiles. Duration of the study will be three years.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who report a physician-made diagnosis of asthma
* Non-smokers and ex-smokers (should have stopped smoking at least 1 year ago)

Exclusion Criteria:

* Contraindications to exercise
* Inability to exercise
* Current smokers or those who stopped smoking within the last week
* Presence of other lung diseases besides asthma
* Patients on systemic steroids
* Major co-morbidities inhibiting participants from being involved in an exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Post-bronchodilator Forced Expired Volume in one second (FEV1) | At baseline (pre-exercise) and two different time points (3 and 6 months of post-exercise)
  Investigators are expecting positive changes (improvement) in Forced Expired Volume in one second (FEV1) over the course of time. FEV1 is an indicator of improvement in the lung functions and, therefore, asthma control.

SECONDARY OUTCOMES:
Improvement in other pulmonary functions as well as quality of life assessment | At baseline (pre-exercise) and two different time points (3 and 6 months of post-exercise)
  Other pulmonary function tests will be measured for the assessment of pulmonary function. A standard Asthma Control Questionnaire will be used to measure improvement in the quality of life
Change in Fraction of exhaled nitric oxide (FeNO) | At baseline (pre-exercise) and two diiferent time points (3 and 6 months of post-exercise)
Change in Immunological Markers | At baseline (pre-exercise) and two different time points (3 and 6 months of post-exercise)
  To determine how the protocol specific intervention affects Immunological Markers.

CONTACTS AND LOCATIONS:
Overall Officials: Rasheed Ahmad, PhD, Principal Investigator — Principal Investigator, Dasman Diabetes Institute; Fahad Al-Ghimlas, MD, Principal Investigator — Co-Principal Investigator, Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No